CLINICAL TRIAL: NCT06134336
Title: The Effect of Eating Disorder on Occupational Balance in University Students
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Busra Kaplan Kilic, Lecturer, Ankara Medipol University
Other Study IDs: 2023/142
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: University Student; Eating Disorders; Occupational Balance
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Research Group: Participants with eating disorders according to the SCOFF Eating Disorders Scale will constitute the research group. Both groups will complete the Occupational Balance Questionnaire and their occupational balances will be compared. The study will be terminated when there are at least 105 participants in the research and control groups and 210 participants in total.
  Interventions: Other: Interview
- Control Group: Participants without eating disorders according to the SCOFF Eating Disorders Scale will constitute the control group. Both groups will complete the Occupational Balance Questionnaire and their occupational balances will be compared. The study will be terminated when there are at least 105 participants in the research and control groups and 210 participants in total.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — No interventional or behavioral intervention will be applied. Only interviews will be conducted through a questionnaire.

SUMMARY:
The aim of this study is to examine the effect of eating disorders on occupational balance in university students. Occupational balance levels will be compared in university students with and without eating disorders. The study will be finalized with the voluntary participation of 105 university students for both groups and 210 university students in total. The relationship between eating disorder tendencies and occupational balance in university students will be examined.

DETAILED DESCRIPTION:
The population of the study will consist of voluntary students between the ages of 18-25 who continue their university education. In the power analysis performed to determine the sample size, it was determined in the G*Power program, with 95% power (alpha = .05, two-way), the effect size was taken as Cohen's d = 0.5 by the guidelines provided by J. Cohen, and it was determined that at least 105 people in each group and 210 people in total were needed for the independent sample t-test.

Inclusion criteria:

* Volunteering to participate in the study,
* To be able to read and write Turkish,
* To be between the ages of 18-25 and studying at undergraduate level

Exclusion criteria:

* Any disability,
* Presence of a chronic disease

Individuals who volunteered to participate in the study will be evaluated with data collection forms filled in through questionnaires. Demographic information about the individuals (such as class, department, age, and gender) will be obtained with the sociodemographic information form. Data collection tools will be used by the researchers in face-to-face interviews with the participants and the data will be recorded anonymously.

It will be determined whether the participants have an eating disorder according to the results of the SCOFF Eating Disorders Scale. Participants with eating disorders will constitute the research group and participants without eating disorders will constitute the control group. Both groups will complete the Occupational Balance Questionnaire and their occupational balances will be compared. The study was planned to be terminated when there were at least 105 participants in each of the research and control groups for the endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* To be able to read and write Turkish,
* To be between the ages of 18-25 and studying at undergraduate level.

Exclusion Criteria:

* Having any disability,
* Presence of a chronic disease.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of the study will consist of volunteer students between the ages of 18-25 who continue their university education.
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
SCOFF Eating Disorders Scale | 5 minute
  The SCOFF Eating Disorders Scale will be used to measure whether the participants have an eating disorder. The Turkish validity and reliability of this scale in university students was conducted by Aydemir et al. in 2015. There are five questions in the scale and the questions are answered as yes/no. One point is given for each question answered as yes, and scores of 2 and above are considered as eating disorders. This scale will be decisive in the inclusion of the participants in the research and control groups.

SECONDARY OUTCOMES:
Occupational Balance Questionnaire | 8 minute
  The Occupational Balance Questionnaire will be used to measure the occupational balance of individuals. This scale defines the concept of occupational balance by measuring the individual's satisfaction with the number and type of activities of daily living. Each item in the scale is a four-point Likert scale ranging from "strongly agree (0)", "disagree (1)", "agree (2)" and "strongly agree (3)". The scores of all items are summed and written as a total score. Scores that can be obtained in the scale vary between 0-33. A high score is characterized as good occupational balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Phillips L, Kemppainen JK, Mechling BM, MacKain S, Kim-Godwin Y, Leopard L. Eating disorders and spirituality in college students. J Psychosoc Nurs Ment Health Serv. 2015 Jan;53(1):30-7. doi: 10.3928/02793695-20141201-01. Epub 2014 Dec 10. PMID 25490775
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25490775/

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT06134336/Prot_ICF_000.pdf